CLINICAL TRIAL: NCT00543140
Title: A Post Implantation/Post Market Evaluation of Safety and Quality of Life in Subjects Implanted With the Swedish Adjustable Gastric Band (SAGB) During Protocol CI-02-0006
Brief Title: Post Implantation/Post Market Evaluation of the Swedish Adjustable Gastric Band
Acronym: SAGB-PM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ethicon Endo-Surgery (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CI-06-0001/CI-07-0006; NCT00813462 (obsolete NCT alias)
Record Dates: First submitted 2007-08-28; First posted 2007-10-12 (Estimated); Results first posted 2016-03-09 (Estimated); Last update posted 2016-03-09 (Estimated); Status verified 2016-02

CONDITIONS: Morbid Obesity
Keywords: Obesity; Morbid Obesity
MeSH Terms: conditions — Obesity, Morbid; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- REALIZE™ Swedish Adjustable Gastric Band (Other): All subjects have the REALIZE™ Swedish Adjustable Gastric Band. Single arm - no comparator.
  Interventions: Device: REALIZE™ Swedish Adjustable Gastric Band

INTERVENTIONS:
Device: REALIZE™ Swedish Adjustable Gastric Band — Laparoscopic placement of the Swedish Adjustable Gastric Band
  Other Names: REALIZE Band

SUMMARY:
The purpose of the study is to evaluate the long term safety of the Swedish Adjustable Gastric Band (SAGB) in subjects with an SAGB in place. Specifically it is designed to determine the re-operation rate (band revision, band replacement and explants resulting from serious adverse device-related event {SADE}) of gastric banding at 4 and 5 year post implant.

DETAILED DESCRIPTION:
NCT00543140 (CI-06-0001) is the 2 year Safety and QOL subject follow-up study to NCT00166205 (CI-02-0006), completed on November 10, 2008. As a condition of approval, the FDA required additional subjects with long-term safety data. These subjects enrolled under protocol CI-07-0006 (NCT00813462)-5 Year Post-Approval Study With the REALIZE (TM) Adjustable Gastric Band. Protocol CI-06-0001 was amended to combine these study subjects with study subjects from CI-07-0006. NCT00543140 (CI-06-0001) will not be completed (analysis of results) until the additional subjects in NCT00813462 (CI-07-0006) complete this study since the original intent was to pool the data together from the above two studies to obtain the appropriate sample size for estimation of the re-operation rate at 4 and 5 years post implantation.

ELIGIBILITY:
CI-06-0001 Inclusion Criteria:

Subjects eligible to participate in this study must fulfill all of the following criteria:

1. Able to comprehend, follow and give signed informed consent;
2. Consented to, and participated in EES Protocol CI-02-0006 titled "A Single-Arm, Multi-Center Study of the Safety and Effectiveness of The Swedish Adjustable Gastric Band (SAGB) in the Treatment of Morbid Obesity";
3. Currently have an SAGB implant in place;
4. Able to commit to long-term follow-up; up to 5 years after SAGB implantation, including band adjustment visits; and
5. Living within the contiguous U.S.

CI-07-0006 Inclusion Criteria:

Subjects eligible to participate in this study must fulfill all of the following criteria:

1. Able to comprehend, follow and give informed consent;
2. 18 to 60 years of age (inclusive);
3. Body Mass Index (BMI) of > 40 kg/m2 and £ 55 kg/m2, or BMI ³ 35 kg/m2 and < 40 kg/m2 with one or more co-morbid conditions.
4. Candidate for surgical weight loss intervention in accordance with the Instructions For Use (i.e., meets acceptable health criteria for major surgery).

CI-06-0001 Exclusion Criteria:

Subjects with the following are not eligible to participate in this clinical trial and must not be enrolled in this study:

a. Consented to, and participated in EES Protocol CI-02-0006 titled "A aSingle-Arm, Multi-Center Study of the Safety and Effectiveness of The Swedish Adjustable Gastric Band (SAGB) in the Treatment of Morbid Obesity"; and have had the SAGB explanted.

CI-07-0006 Exclusion Criteria:

1. Women who are currently pregnant.
2. Previous malabsorptive or restrictive procedures performed for the treatment of morbid obesity.
3. Documented history of drug and/or alcohol abuse within 2 years of the Screening Visit (1a).
4. Presence of any of the following medical conditions;

   1. Inflammatory diseases of the gastrointestinal tract, including severe intractable esophagitis, gastric ulceration or duodenal ulceration, or specific inflammation such as Crohn's disease;
   2. Severe cardiopulmonary disease or other serious organic disease;
   3. Upper gastrointestinal bleeding conditions such as esophageal or gastric varices or intestinal telangiectases;
   4. Portal hypertension;
   5. Anomalies of the gastrointestinal tract such as atresia or stenosis;
   6. Cirrhosis of the liver;
   7. Chronic pancreatitis;
   8. Patients on chronic, long-term steroid treatment or steroids within 15 days of surgery;
   9. Unable or unwilling to comply with dietary restrictions required by this procedure;
   10. Known allergy to materials contained within the band or its injection port (silicone elastomer containing 10% BaSO4, polyetheretherketone (PEEK), and cobalt chromium)
5. Presence of terminal illness with life expectancy of £ 5 years.
6. Inability to refrain from use of anticoagulants or aspirin within 15 days prior to surgery.
7. Acute or chronic infection (localized or systemic).
8. Participation in another clinical trial within 8 weeks of the Screening Visit (1a) and for the duration of this trial.
9. Any medical condition or finding for which the Investigator utilizes their medical discretion to determine the subject should be excluded due to inability to understand or follow study procedures.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 303 (Actual)
Dates: Start 2006-08; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward Phillips, MD, Principal Investigator — Cedars Sinai
Locations (8):
- United States (8):
  - Surgical Associates of La Jolla Medical Group, Inc., La Jolla, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Advanced Surgical Institute at Mercy Hospital, Miami, Florida
  - Robert T. Marema, MD, Saint Augustine, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - Hamilton Medical Center - Weight Management, Dalton, Georgia
  - St. Luke's Roosevelt Hospital Center, New York, New York
  - dgd Research, Inc., San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD. Cumulative data from the study will be published.

RESULTS

PARTICIPANT FLOW:
Groups:
- REALIZE™ Adjustable Gastric Band: All subjects have the REALIZE™ Adjustable Gastric Band. Single arm - no comparator.
  Swedish Adjustable Gastric Band: Laparoscopic placement of the Swedish Adjustable Gastric Band
Period: Overall Study
Arm/Group | REALIZE™ Adjustable Gastric Band
Started | 303
Completed | 231
Not Completed | 72
Not completed — Lost to Follow-up | 33
Not completed — Withdrawal by Subject | 13
Not completed — Protocol Violation | 10
Not completed — Insufficient weight loss | 10
Not completed — SAE leading to explant of SAGB | 3
Not completed — Death | 1
Not completed — Subject moved | 1
Not completed — Conversion to different procedure | 1

BASELINE CHARACTERISTICS:
Population: All subjects implanted with the SAGB.
Arm/Group | REALIZE™ Adjustable Gastric Band
Number analyzed (Participants) | 303
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.5 (9.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 242
  Male | 61
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian, not of Hispanic origin | 205
  Hispanic | 55
  Black, not of Hispanic origin | 27
  Asian/Pacific Islander | 8
  Other | 8
Region of Enrollment [Number; unit: participants]
  United States | 303
Weight (lbs) [Mean (Standard Deviation); unit: pounds] | 272.2 (40.78)
Body Mass Index (kg/m^2) [Mean (Standard Deviation); unit: kilograms per meters squared] | 44.1 (4.76)

OUTCOME MEASURES:

1. Primary Outcome: Re-operation Rate (Band Revision, Band Replacement and Explants Resulting From Serious Adverse Device-related Event {SADE}) of Gastric Banding at 4 and 5 Years Post Implant.
Description: A reoperation was identified by satisfying all of the following criteria:
  * Is an SAE or is the action taken as the result of an SAE;
  * Is related to the device (i.e., has a relationship to study device that is indicated as Definite, Probable, Possible, or Unknown). In cases where the reoperation is the action taken for an SAE, then the SAE itself should be related to the device;
  * Is an explant, band revision, or band replacement resulting from a medical condition (perceived failure of weight loss, subject request, and other non-medical conditions will not be counted); and
  * Has a start date that is strictly more than 1095 days (3 years) from the implantation of the device.
Time Frame: 5 years
Population: Consists of subjects who had a device implanted under protocol CI-07-0006 and subjects implanted under protocol CI-02-0006 and subsequently enrolled under protocol CI-06-0001.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | REALIZE™ Adjustable Gastric Band
Number analyzed (Participants) | 303
percentage of subjects | 8.91 [5.95 to 12.70]
Statistical Analysis 1: Comparison: REALIZE™ Adjustable Gastric Band; The primary analysis used a one-sided binomial exact test method by Clopper and Pearson to determine if the rate of reoperations observed in Years 4 and 5 (combined) of the study was significantly less than 8%. The null hypothesis was that the reoperation rate was greater than or equal to 8%; Test type: Superiority or Other; p = 0.6919, Exact Binomial method — No adjustments for multiple comparisons were performed as only one hypothesis was tested in this study. The level of significance was set at 0.05

2. Secondary Outcome: Change in Glycosylated Hemoglobin (HbA1c) at 5 Years Post Implant.
Description: The natural unit of measurement for HbA1c is percent (%). Results provided represent change from baseline, that is, Year 5 value minus Baseline value.
Time Frame: 5 years
Population: All subjects providing a measurement at the 5 year visit. No imputation of missing data was performed.
Measure: Mean (95% Confidence Interval); unit: percentage
Arm/Group | REALIZE™ Adjustable Gastric Band
Number analyzed (Participants) | 227
percentage | -0.22 [-0.33 to -0.11]

3. Secondary Outcome: Percent Change in Excess Body Weight at 5 Years Post-implant
Time Frame: 5 years
Population: All subjects providing a measurement at the 5 year visit. No imputation of missing data was performed.
Measure: Mean (95% Confidence Interval); unit: percentage of excess body weight
Arm/Group | REALIZE™ Adjustable Gastric Band
Number analyzed (Participants) | 240
percentage of excess body weight | -35.6 [-39.0 to -32.2]

4. Secondary Outcome: Change in SF-36 Health Survey Physical Component at 5 Years Post Implant
Description: Scores on the SF-36 Health Survey are determined by methodology publised with the validated instrument. Scores can range from 0 to 100 with higher scores indicating higher quality of life.
Time Frame: 5 years
Population: All subjects providing a measurement at the 5 year visit. No imputation of missing data was performed.
Measure: Mean (95% Confidence Interval); unit: unitless scale ranging 0 to 100
Arm/Group | REALIZE™ Adjustable Gastric Band
Number analyzed (Participants) | 233
unitless scale ranging 0 to 100 | 8.1 [6.6 to 9.5]

5. Secondary Outcome: Change in SF-36 Health Survey Mental Component at 5 Years Post Implant
Description: as for outcome 4
Time Frame: 5 years
Population: All subjects providing a measurement at the 5 year visit. No imputation of missing data was performed.
Measure: Mean (95% Confidence Interval); unit: Unitless scale ranging 0 to 100
Arm/Group | REALIZE™ Adjustable Gastric Band
Number analyzed (Participants) | 233
Unitless scale ranging 0 to 100 | 1.1 [-0.4 to 2.6]

ADVERSE EVENTS:
Time Frame: Date of Surgery Through 5 Years Post Implantation
Arm/Group | REALIZE™ Adjustable Gastric Band
Serious Adverse Events (participants affected / at risk) | 138/303
Other Adverse Events (participants affected / at risk) | 302/303
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | REALIZE™ Adjustable Gastric Band (N=303)
ANAEMIA (Blood and lymphatic system disorders) | 1 (1)
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 1 (1)
ATRIAL FIBRILLATION (Cardiac disorders) | 3 (3)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1)
BRADYCARDIA (Cardiac disorders) | 1 (1)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 1 (1)
VERTIGO (Ear and labyrinth disorders) | 1 (1)
GASTRIC DILATATION (Gastrointestinal disorders) | 7 (7)
HIATUS HERNIA (Gastrointestinal disorders) | 5 (5)
VOMITING (Gastrointestinal disorders) | 5 (5)
ABDOMINAL PAIN (Gastrointestinal disorders) | 3 (3)
OBSTRUCTION GASTRIC (Gastrointestinal disorders) | 3 (3)
CONSTIPATION (Gastrointestinal disorders) | 2 (2)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 2 (2)
ABDOMINAL ADHESIONS (Gastrointestinal disorders) | 1 (1)
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 1 (1)
DIVERTICULAR PERFORATION (Gastrointestinal disorders) | 1 (1)
DYSPHAGIA (Gastrointestinal disorders) | 1 (1)
GASTRIC ULCER (Gastrointestinal disorders) | 1 (1)
GASTRITIS (Gastrointestinal disorders) | 1 (1)
GASTRITIS EROSIVE (Gastrointestinal disorders) | 1 (1)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1)
GASTROINTESTINAL OEDEMA (Gastrointestinal disorders) | 1 (1)
HAEMORRHOIDS (Gastrointestinal disorders) | 1 (1)
IMPAIRED GASTRIC EMPTYING (Gastrointestinal disorders) | 1 (1)
INTESTINAL PERFORATION (Gastrointestinal disorders) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 1 (1)
OESOPHAGEAL DISORDER (Gastrointestinal disorders) | 1 (1)
OESOPHAGEAL OBSTRUCTION (Gastrointestinal disorders) | 1 (1)
OESOPHAGITIS (Gastrointestinal disorders) | 1 (1)
PEPTIC ULCER (Gastrointestinal disorders) | 1 (1)
REGURGITATION (Gastrointestinal disorders) | 1 (1)
UMBILICAL HERNIA (Gastrointestinal disorders) | 1 (1)
VOLVULUS (Gastrointestinal disorders) | 1 (1)
CATHETER RELATED COMPLICATION (General disorders) | 15 (16)
CHEST PAIN (General disorders) | 4 (4)
IMPLANT SITE PAIN (General disorders) | 2 (2)
ASTHENIA (General disorders) | 1 (1)
DRUG WITHDRAWAL SYNDROME (General disorders) | 1 (1)
IMPLANT SITE HAEMATOMA (General disorders) | 1 (1)
NON-CARDIAC CHEST PAIN (General disorders) | 1 (1)
PYREXIA (General disorders) | 1 (1)
CHOLELITHIASIS (Hepatobiliary disorders) | 13 (13)
CHOLECYSTITIS (Hepatobiliary disorders) | 8 (9)
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 3 (3)
BILIARY DYSKINESIA (Hepatobiliary disorders) | 1 (1)
HEPATIC LESION (Hepatobiliary disorders) | 1 (1)
GRAFT VERSUS HOST DISEASE (Immune system disorders) | 1 (2)
DEVICE RELATED INFECTION (Infections and infestations) | 3 (3)
OSTEOMYELITIS (Infections and infestations) | 3 (3)
PNEUMONIA (Infections and infestations) | 3 (4)
GASTROENTERITIS (Infections and infestations) | 2 (2)
IMPLANT SITE INFECTION (Infections and infestations) | 2 (2)
ABDOMINAL ABSCESS (Infections and infestations) | 1 (1)
ABSCESS (Infections and infestations) | 1 (1)
APPENDICEAL ABSCESS (Infections and infestations) | 1 (1)
APPENDICITIS (Infections and infestations) | 1 (1)
BACTERIAL PYELONEPHRITIS (Infections and infestations) | 1 (1)
BRONCHITIS (Infections and infestations) | 1 (1)
KIDNEY INFECTION (Infections and infestations) | 1 (1)
POSTOPERATIVE ABSCESS (Infections and infestations) | 1 (1)
RENAL ABSCESS (Infections and infestations) | 1 (1)
STAPHYLOCOCCAL BACTERAEMIA (Infections and infestations) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1)
DEVICE MIGRATION (Injury, poisoning and procedural complications) | 28 (31)
DEVICE FAILURE (Injury, poisoning and procedural complications) | 5 (5)
DEVICE MALFUNCTION (Injury, poisoning and procedural complications) | 3 (3)
FOOT FRACTURE (Injury, poisoning and procedural complications) | 2 (2)
PROCEDURAL COMPLICATION (Injury, poisoning and procedural complications) | 2 (2)
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 2 (2)
DEVICE OCCLUSION (Injury, poisoning and procedural complications) | 1 (1)
FACIAL BONES FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
FAILURE OF IMPLANT (Injury, poisoning and procedural complications) | 1 (1)
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
INJURY (Injury, poisoning and procedural complications) | 1 (1)
LIGAMENT INJURY (Injury, poisoning and procedural complications) | 1 (1)
MENISCUS LESION (Injury, poisoning and procedural complications) | 1 (1)
OVERDOSE (Injury, poisoning and procedural complications) | 1 (1)
WOUND DEHISCENCE (Injury, poisoning and procedural complications) | 1 (1)
DEHYDRATION (Metabolism and nutrition disorders) | 1 (2)
FOOD INTOLERANCE (Metabolism and nutrition disorders) | 1 (1)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 (1)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 6 (6)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2 (2)
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 2 (2)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (1)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1)
INTERVERTEBRAL DISC DISORDER (Musculoskeletal and connective tissue disorders) | 1 (1)
LUMBAR SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 1 (1)
PLANTAR FASCIITIS (Musculoskeletal and connective tissue disorders) | 1 (1)
ROTATOR CUFF SYNDROME (Musculoskeletal and connective tissue disorders) | 1 (1)
SCOLIOSIS (Musculoskeletal and connective tissue disorders) | 1 (1)
UTERINE LEIOMYOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
ACUTE MYELOID LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
BENIGN BREAST NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
BRAIN NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
BENIGN INTRACRANIAL HYPERTENSION (Nervous system disorders) | 1 (1)
HEADACHE (Nervous system disorders) | 1 (2)
INTRACRANIAL PRESSURE INCREASED (Nervous system disorders) | 1 (1)
ANXIETY (Psychiatric disorders) | 1 (2)
PSYCHOTIC DISORDER (Psychiatric disorders) | 1 (1)
SUICIDAL IDEATION (Psychiatric disorders) | 1 (1)
NEPHROLITHIASIS (Renal and urinary disorders) | 1 (1)
RENAL FAILURE ACUTE (Renal and urinary disorders) | 1 (1)
URINARY RETENTION (Renal and urinary disorders) | 1 (1)
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 1 (1)
CERVICAL DYSPLASIA (Reproductive system and breast disorders) | 1 (1)
ENDOMETRIAL HYPERPLASIA (Reproductive system and breast disorders) | 1 (1)
MENORRHAGIA (Reproductive system and breast disorders) | 1 (1)
OVARIAN CYST (Reproductive system and breast disorders) | 1 (1)
POSTMENOPAUSAL HAEMORRHAGE (Reproductive system and breast disorders) | 1 (1)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 2 (2)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 2 (2)
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 1 (1)
SKIN DISORDER (Skin and subcutaneous tissue disorders) | 1 (1)
COLOSTOMY (Surgical and medical procedures) | 1 (1)
MEDICAL DEVICE CHANGE (Surgical and medical procedures) | 1 (1)
DEEP VEIN THROMBOSIS (Vascular disorders) | 3 (3)
THROMBOSIS (Vascular disorders) | 2 (2)
HYPOTENSION (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | REALIZE™ Adjustable Gastric Band (N=303)
ANAEMIA (Blood and lymphatic system disorders) | 17 (18)
VOMITING (Gastrointestinal disorders) | 188 (547)
NAUSEA (Gastrointestinal disorders) | 113 (181)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 87 (140)
CONSTIPATION (Gastrointestinal disorders) | 85 (106)
DYSPEPSIA (Gastrointestinal disorders) | 78 (126)
DYSPHAGIA (Gastrointestinal disorders) | 68 (91)
ABDOMINAL PAIN (Gastrointestinal disorders) | 52 (57)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 47 (59)
OESOPHAGEAL DILATATION (Gastrointestinal disorders) | 42 (49)
HIATUS HERNIA (Gastrointestinal disorders) | 36 (40)
FLATULENCE (Gastrointestinal disorders) | 35 (38)
DIARRHOEA (Gastrointestinal disorders) | 28 (39)
GASTRIC DILATATION (Gastrointestinal disorders) | 26 (28)
FATIGUE (General disorders) | 33 (41)
IMPLANT SITE PAIN (General disorders) | 33 (33)
PYREXIA (General disorders) | 23 (33)
OEDEMA PERIPHERAL (General disorders) | 18 (21)
CHEST PAIN (General disorders) | 17 (19)
SEASONAL ALLERGY (Immune system disorders) | 17 (18)
NASOPHARYNGITIS (Infections and infestations) | 63 (103)
SINUSITIS (Infections and infestations) | 48 (75)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 42 (52)
URINARY TRACT INFECTION (Infections and infestations) | 42 (59)
INFLUENZA (Infections and infestations) | 35 (42)
GASTROENTERITIS VIRAL (Infections and infestations) | 31 (38)
BRONCHITIS (Infections and infestations) | 25 (30)
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 176 (227)
PROCEDURAL NAUSEA (Injury, poisoning and procedural complications) | 48 (49)
BLOOD CHOLESTEROL INCREASED (Investigations) | 25 (27)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 37 (45)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 35 (42)
HEADACHE (Nervous system disorders) | 43 (48)
DEPRESSION (Psychiatric disorders) | 37 (41)
INSOMNIA (Psychiatric disorders) | 34 (41)
ANXIETY (Psychiatric disorders) | 28 (33)
COUGH (Respiratory, thoracic and mediastinal disorders) | 16 (16)
ALOPECIA (Skin and subcutaneous tissue disorders) | 42 (46)
HYPERTENSION (Vascular disorders) | 53 (62)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PIs agreed that the first publication of results should be made in conjunction with the presentation of a joint, multicenter publication of the results with the PIs from all sites contributing data, analyses, and comments. If this publication was not submitted within 12 months after conclusion of the Study at all sites, or after Sponsor confirmed there would be no multicenter Study publication, whichever is first, the PIs could have published the results from their individual sites.